CLINICAL TRIAL: NCT07160842
Title: Impact of a School-based Educational Intervention That Combined a Structured Training Session With a Fluorescence-enabled Device on the Quality of Students' Hand Hygiene at 1, 3 and 6 Months Post Intervention
Brief Title: Impact of an AI-enabled UV Hand Hygiene Intervention in Primary Schools: a Community Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Catala de Salut (Other Government)
Collaborators: CEEISCAT (Unknown); Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Principal Investigator, Anna Bordas, Doctor in Pharmacology, Institut Catala de Salut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Handhygiene_sentinelschools
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Intervention in Hand Hygiene for Infectious Diseases Prevention
Keywords: hand hygiene; prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The educational intervention consisted of a two-part training session: (i) a thirty-minute didactic session introducing the 7-step alcohol-based hand rub (ABHR) technique (14), the importance of proper hand hygiene for infection prevention; and (ii) a practical component on hand hygiene with real-time feedback
  Interventions: Behavioral: Hand hygiene intervention
- Control group (No Intervention): The control group received the hand hygiene evaluation visits without the educational session

INTERVENTIONS:
Behavioral: Hand hygiene intervention — The educational intervention consisted of a two-part training session: (i) a thirty-minute didactic session introducing the 7-step alcohol-based hand rub (ABHR) technique (14), the importance of proper hand hygiene for infection prevention; and (ii) a practical component on hand hygiene with real-time feedback.
  Arms: Intervention group

SUMMARY:
Background Hand hygiene refers to the practice of keeping hands clean to prevent the spread of disease. Hand hygiene workshops are an important tool to educate students about the importance of keeping their hands clean and healthy.

Objectives The primary objective of this project is to evaluate the effectiveness of an educational intervention previously used in other settings that incorporates a fluorescence-based device to quantify the quality of hand hygiene in real time, together with a training workshop for students, with the aim of improving health promotion and prevention in the short and medium term (1, 3, and 6 months).

Methods This is a sub-study of the Sentinel Schools Project. It is a controlled before-after study with school level allocation using a single matched pair (1 intervention school; 1 control school) and repeated measures conducted in schools belonging to the Sentinel Schools network within the Camp de Tarragona health region. The study population comprises students enrolled in primary education at these schools. The project field team carried out a pre-intervention assessment of handwashing quality in both study arms using a device that uses fluorescence to detect adequately washed areas of the hand. In the intervention arm, an educational training session on hand hygiene was delivered, followed by post-intervention assessments at short and medium term in both study arms. To examine the acceptability of the intervention, an ad hoc questionnaire was administered to the teachers who supervise the participating classes and also focal groups and enterprises were made to access the acceptability of the intervention.

Statistical Analysis Frequencies and percentages will be calculated for qualitative variables; for quantitative variables, the mean and standard deviation, as well as minimum and maximum values, will be reported. Ninety-five percent confidence intervals will be presented for means and for proportions. Bivariate analyses for quantitative variables will be performed, estimating Pearson correlation coefficients and/or linear regression.

ELIGIBILITY:
Inclusion Criteria:

* students attending third- to sixth-grade of enrolled primary school

Exclusion Criteria:

* physical or intellectual disabilities precluding correct hand hygiene
* allergy/contraindication to alcohol-based hand rub (ABHR)
* <80% school attendance.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2024-03-02 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Percentage of hand surface area correctly washed | From enrollment to the end of the evaluation visits at 6 months
  The percentage of clean hand surface area, defined as the proportion of the total hand that was adequately covered with hand rub

CONTACTS AND LOCATIONS:
Locations (1):
- Cap Sant Pere, Reus, Spain

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared. This trial was conducted in schools with minors, and informed consent did not include permission to share de-identified IPD beyond the study team. In alignment with ethical approvals and applicable data protection regulations, only aggregate results will be made publicly available.